CLINICAL TRIAL: NCT02010892
Title: Effective Treatments for Thoracic Aortic Aneurysms (ETTAA Study): A Prospective Cohort Study
Acronym: ETTAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: P01633; 11/147/03 (Other Grant/Funding Number: NIHR Health Technology Assessment Programme)
Record Dates: First submitted 2013-11-22; First posted 2013-12-13 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic | interventions — Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Watchful Waiting: Patients with aneurysms considered to be at low risk of rupture will remain under surveillance with annual CT / MRI scans and multi-disciplinary team review (as per local practice). These patients' data will contribute to the natural history component of the study.
- Best Medical Therapy: This refers to lifestyle modification (smoking cessation and dietary management) as well as medical management of hypercholesterolaemia and hypertension for patients who are considered unsuitable for, or who refuse, OSR / ESG.
- Open Surgery (OSR): Replacement of the aneurysmal aorta with prosthetic conduit via a sternotomy or thoracotomy with circulatory support.
  Interventions: Procedure: Open Surgery (OSR)
- Stenting (ESR): Endovascular repair of the aneurysm via transluminal introduction of a stent-graft under X-ray guidance. Hybrid procedures that comprise a combination of a conventional surgical component and a transluminal repair are to be included in this group.
  Interventions: Procedure: Stent Grafting (ESR)

INTERVENTIONS:
Procedure: Stent Grafting (ESR)
  Groups: Stenting (ESR)
Procedure: Open Surgery (OSR)
  Groups: Open Surgery (OSR)

SUMMARY:
This is a prospective observational cohort study that will collect data from the point of referral through to secondary care, aiming for 3 years median follow-up (range 1-5 years). The data collected will allow estimation of the success of any intervention (in terms of reducing rate of aneurysm growth, rupture or dissection) as well as estimation of the risks associated with the three procedures. Clinical outcomes in the three treatment groups will be described.

Aims

We aim to answer the following questions:

1. Without procedural intervention for chronic thoracic aortic aneurysm (CTAA), what is the risk of aneurysm growth, dissection, rupture, permanent neurological injury or death? What is the effect on quality of life (QoL)?
2. If a patient has endovascular stent grafting (ESG) or open surgical repair (OSR), what is the risk of growth, dissection, rupture, permanent neurological injury or death?
3. How does QoL change from pre- to post intervention?
4. Can aneurysm or patient related predictors of good/poor treatment outcomes be determined?
5. What is the most cost-effective strategy in:

   1. Patients eligible for either ESG or OSR?
   2. Patients eligible for either ESG or best medical therapy (BMT)?
   3. Patients eligible for either watchful waiting (WW) or intervention (ESG/ OSR)?
6. What further research is required? What would be the most important research to pursue?

ELIGIBILITY:
Inclusion Criteria:

* Thoracic Aortic Aneurysm > 4cm
* Age ≥18 years
* Able to give informed consent

Exclusion Criteria:

* Intervention required below the level of the coeliac axis
* Acute dissection or malperfusion syndromes (such as myocardial infarction,acute stroke or limb ischaemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being referred to a specialist centre for diagnosis and treatment of their aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Aneurysm Growth | 1, 2, 3 , 4 and 5 years post recruitment
Quality of life | 1, 2, 3 , 4 and 5 years post recruitment
Freedom from reintervention | 1, 2, 3 , 4 and 5 years post recruitment
Freedom from death or permanent neurological injury | 1, 2, 3 , 4 and 5 years post recruitment
Costs to the NHS | 1, 2, 3 , 4 and 5 years post recruitment
Incremental cost per quality adjusted life year gained | 1, 2, 3 , 4 and 5 years post recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Large, FRCS, Study Chair — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Cambridge, Cambs, United Kingdom

REFERENCES:
- [Derived] Sharples L, Sastry P, Freeman C, Gray J, McCarthy A, Chiu YD, Bicknell C, McMeekin P, Vallabhaneni SR, Cook A, Vale L, Large S. Endovascular stent grafting and open surgical replacement for chronic thoracic aortic aneurysms: a systematic review and prospective cohort study. Health Technol Assess. 2022 Jan;26(6):1-166. doi: 10.3310/ABUT7744. PMID 35094747